CLINICAL TRIAL: NCT05446636
Title: Circadian Rhythm Status and CS (Cesarean Section) Postoperative Pain
Status: Recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Biological rhythm and CS pain
Record Dates: First submitted 2022-06-01; First posted 2022-07-07 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-06

CONDITIONS: Circadian Rhythm
Keywords: Circadian Rhythm; Cesarean Section; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Huawei bracelet — Huawei bracelet was used to continuously record maternal respiration, heart rate, temperature and sleep data, and then calculate maternal circadian rhythm state

SUMMARY:
Use huawei wristwatch to record maternal rhythm status and record the VAS score after cesarean section under combined spinal-epidural anesthesia. Based on this study the investigators intend to explore the correlation between maternal circadian rhythm status and postoperative pain after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 45
* ASA(American society of anesthesiologists) status II-III
* 37-42 weeks gestation
* undergo elective cesarean section with subarachnoid anesthesia
* participate in this study and sign informed consent

Exclusion Criteria:

* Patients with contraindications of combined spinal and epidural anesthesia
* Patients with severe systemic disease
* Alcoholism and long-term use of anti-inflammatory and analgesic drugs
* Patients who were unable to cooperate or refused to participate in the trial
* with psychiatric disorder
* researchers considered unsuitable to participate in or unable to cooperate with the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate and severe pain after cesarean section | From ending of the surgery to 24hours after cesarean section
  number rating scale (NRS) for pain (0=no pain to 10=worst pain) >4

SECONDARY OUTCOMES:
Pain intensity durig 0 to 6 hours after surgery | From ending of the surgery to 6 hours after cesarean section
  number rating scale (NRS) for pain (0=no pain to 10=worst pain)
Pain intensity durig 6 to 12 hours after surgery | From 6 hours after cesarean section to 12 hours after cesarean section
  number rating scale (NRS) for pain (0=no pain to 10=worst pain)
Pain intensity durig 12 to 24 hours after surgery | From 12 hours after cesarean section to 24 hours after cesarean section
  number rating scale (NRS) for pain (0=no pain to 10=worst pain)
Heart rate variability | From the time of inclusion in the study until the patient's postoperative discharge, assessed up to 1 week
  Heart rate variability recorded by Huawei bracelet
Body temperature variability | From the time of inclusion in the study until the patient's postoperative discharge, assessed up to 1 week
  Body temperature variability recorded by Huawei bracelet
Variability of patients' activity | From the time of inclusion in the study until the patient's postoperative discharge, assessed up to 1 week
  Variability of patients' activity recorded by Huawei bracelet
Percentage of deep sleep | From the time of inclusion in the study until the patient's postoperative discharge, assessed up to 1 week
  Percentage of deep sleep evaluated by Huawei bracelet
Percentage of rapid eye movement sleep | From the time of inclusion in the study until the patient's postoperative discharge, assessed up to 1 week
  Percentage of rapid eye movement sleep evaluated by Huawei bracelet

CONTACTS AND LOCATIONS:
Overall Officials: Guangyou Duan, MD, Study Director — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years